CLINICAL TRIAL: NCT03088644
Title: An Open-label Study to Investigate P2X7 Receptor Occupancy by JNJ-54175446 With the Newly Developed P2X7 Receptor PET Tracer 18F-JNJ-64413739
Brief Title: A Study to Investigate P2X7 Receptor Occupancy by JNJ-54175446 With the Newly Developed P2X7 Receptor Positron Emission Tomography (PET) Tracer 18F-JNJ-64413739
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108269; 2016-004007-31 (EudraCT Number); 54175446EDI1004 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-54175446; (18)F-JNJ-64413739

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: 18F-JNJ-64413739 (Experimental): Subjects will receive an intravenous (IV) bolus injection of 18F-JNJ-64413739 at a dose between 150 and 185 megaBecquerel (MBq) on Day 1 of Part A to investigate the total body biodistribution and measure the radiation dosimetry.
  Interventions: Drug: 18F-JNJ-64413739
- Part B: 18F-JNJ-64413739 (Experimental): Subjects will receive an IV bolus injection of 18F-JNJ-64413739 at a dose between 150 and 185 MBq on Day 1 of Part B to measure the uptake, distribution, and clearance in brain.
  Interventions: Drug: 18F-JNJ-64413739
- Part C: 18F-JNJ-64413739 (Experimental): Subjects will receive an IV bolus injection of 18F-JNJ-64413739 for a PET/MR scan on Day 1 and a repeat 18F-JNJ-64413739 PET/magnetic resonance (MR) scan at least 1 week later to determine the test-retest variability in V[t]. 18F-JNJ-64413739 doses will be between 150 and 185 MBq.
  Interventions: Drug: 18F-JNJ-64413739
- Part D: JNJ-54175446 + 18F-JNJ-64413739 (Experimental): Subjects will have a baseline 18F-JNJ-64413739 PET/MR scan on Day 1. On Day 2 they will receive JNJ-54175446 (maximum 600 milligram [mg]) orally (after light breakfast) and then an IV injection of 18F-JNJ-64413739 four hours after dosing for a PET/MR scan. At least 1 week later, they will receive another dose of JNJ-54175446, and then an IV injection of 18F-JNJ-64413739 four hours later for a second post-treatment PET/MR scan. 18F-JNJ-64413739 doses will be between 150 and 185 MBq.
  Interventions: Drug: JNJ-54175446

INTERVENTIONS:
Drug: JNJ-54175446 — JNJ-54175446 up to 600 mg suspension for oral dose administration.
  Arms: Part D: JNJ-54175446 + 18F-JNJ-64413739
Drug: 18F-JNJ-64413739 — 18F-JNJ-64413739 fluid for injection administered intravenously.
  Arms: Part A: 18F-JNJ-64413739; Part B: 18F-JNJ-64413739; Part C: 18F-JNJ-64413739

SUMMARY:
The primary purpose of this study is to measure the whole body distribution and radiation dosimetry of 18F-JNJ-64413739 (Part A), to measure the uptake, distribution, and clearance (CL) of 18F-JNJ-64413739 in the brain of healthy male subjects by Positron Emission Tomography (PET) and to model tissue specific kinetics of 18F-JNJ-64413739 with the appropriate input function (IF) (Part B), to measure subject test retest variability in the distribution of 18F-JNJ-64413739 in the brain of healthy male subjects by comparing PET scans obtained at least 1 week apart (Part C) and following single oral dose administration of JNJ-54175446, to measure the blocking of 18F-JNJ-64413739 uptake in the brain at the time to reach maximum plasma concentration (tmax) of JNJ-54175446 and model the exposure/receptor interaction of JNJ-54175446 in healthy male subjects (Part D).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) inclusive (BMI = weight/height^2)
* Nonsmoker (not smoked for 3 months prior to screening)
* Is willing to allow the investigators to place an arterial catheter in the radial artery, is assessed via physical examination (Allen Test) to be a good subject for arterial catheter placement and should not be allergic to local anesthetics for catheter placement (Part B-C-D)
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, in addition to the highly effective method of contraception, a man: who is sexually active with a woman of childbearing potential and has not had vasectomy must agree to use a barrier method of contraception (e.g., condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository). In addition, their female partner should also use an highly effective method of birth control (e.g. hormonal contraception) for at least the same duration; who is sexually active with a woman who is pregnant must use a condom; must agree not to donate sperm
* Subjects must have signed an informed consent document indicating that they understand the purpose of, and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Exposed to greater than (>)1 millisievert (mSv) of ionizing radiation participating as a subject in research studies in the 12 months before the start of this study
* Clinically significant abnormal physical and neurological examination, vital signs or 12-lead electrocardiogram (ECG) at screening or admission
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, parkinson's disease, infection, or any other illness that the Investigator considers should exclude the subject. History of epilepsy or fits or unexplained black-outs
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies
* Subject has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 6 months before Screening or positive test result(s) for alcohol and/or drugs of abuse (opiates (including methadone), cocaine, amphetamines, methamphetamines, cannabinoids, barbiturates, ecstasy and benzodiazepines) at screening or admission of each period

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Part A: Effective Radiation Dose Following Injection of 18F-JNJ-64413739 | Up to 4 Weeks
  The tissue radioactivity will be measured per organ for up to 5 hours after injection of up to 185 megaBecquerel (MBq) of 18F-JNJ-64413739 and corrected for attenuation by computed tomography (CT) transmission scans using PET/CT. These measurements will be used to estimate effective radiation dose per organ and total body.
Part B: Total and Regional Brain Compartmental Kinetics for Volume of Distribution of 18F-JNJ-64413739 | Up to 4 Weeks
  The Distribution of 18F-JNJ-64413739 in brain will be measured by dynamic PET/magnetic resonance (MR) scans obtained from the time of injection for up to 120 minutes along with measurement of the tracer input function with arterial samples for intact tracer and metabolites to establish the total and regional compartmental kinetics and volume of distribution (V[t]) of 18F-JNJ-64413739.
Part C: Test Retest Variability in the Distribution of 18F-JNJ-64413739 | Up to 5 Weeks
  Test Retest Variability within subjects will be assessed based on percent difference in V[t] following 18F-JNJ-64413739 PET/MR scans obtained at least 1 Week apart. V[t] will be the parameter for the estimated volume of distribution of the tracer derived from the kinetic model that best fits the data from Part B. It will be calculated by formula [100*abs (V[t]test - V[t]retest)/[( V[t]test+ V[t]retest)/2].
Part D: Plasma Concentrations of JNJ-54175446 | Up to 5 Weeks
  Descriptive statistics will be calculated for the plasma concentrations of JNJ-54175446.
Part D: Percentage of P2X7 Receptor Occupancy | Up to 5 Weeks
  Percent reduction in V[t] of 18F-JNJ-64413739 in brain regions of interest will be calculated by PET/MR scans obtained at pre and post treatment with single doses of JNJ-54175446.

SECONDARY OUTCOMES:
Part A, B and C: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of 18F-JNJ-64413739 | Part A and B: Up to 4 Weeks; Part C: Up to 5 Weeks
  An adverse event is any untoward medical event that occurs in a subject administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part D: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of JNJ-54175446 | Up to 5 Weeks
  An adverse event is any untoward medical event that occurs in a subject administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- UZ Leuven, Leuven, Belgium